CLINICAL TRIAL: NCT06147271
Title: Impact of SGLT2 Inhibitors on Cardioprotection in Patients Undergoing Heart Transplantation
Brief Title: Impact of SGLT2 Inhibitors in Heart Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Collaborators: Hospital de Messejana (Unknown)
Responsible Party: Principal Investigator, Jefferson Luis Vieira, Jefferson Vieira, MD, MBA, PHD, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SGLT2i and heart transplant
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Transplant; Failure, Heart; Cardiac Allograft Vasculopathy; Rejection Heart Transplant
Keywords: heart transplantation; Cardiac Allograft Vasculopathy; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): All adult patients undergoing a heart transplant between January 2017 and December 2023 at Hospital de Messejana randomized to SGLT2i intervention
  Interventions: Drug: SGLT2i
- no intervention (No Intervention): All adult patients undergoing a heart transplant between January 2017 and December 2023 at Hospital de Messejana randomized to routine surveillance

INTERVENTIONS:
Drug: SGLT2i — A randomized clinical trial of superiority with active control (2 arms), with central randomization to evaluate the efficacy and safety of adding dapagliflozin or empagliflozin 10 mg once daily to post-TxC routine compared with no intervention for 6-8 months.
  Arms: intervention

SUMMARY:
The goal of this clinical trial is to test if SGLT2 inhibitors could prevent or delay the development of Cardiac Allograft Vasculopathy (CAV) post-heart transplantation (TxC). The main questions it aims to answer are:

Primary outcome: CAV, according to ISHLT grading system diagnosed by CCTA; Secondary outcomes: cardiovascular death, all-cause mortality, hospitalization, worsening glomerular filtration rate, fasting glucose, weight, and blood pressure.

Exploratory and safety outcomes: Rejection, hypoglycemia, urinary tract infection, hypovolemia, and limb amputation.

HYPOTHESIS The null hypothesis is that SGLT2 inhibitors do not reduce the incidence of CAV in transplanted patients.

The alternative hypothesis is that SGLT2 inhibitors reduce the incidence of CAV in transplanted patients.METHODOLOGY Study Design A randomized clinical trial of superiority with active control (2 arms), with central randomization and blinded evaluation of outcomes, to evaluate the efficacy and safety of adding dapagliflozin or empagliflozin 10 mg once daily to conventional post-TxC treatment compared with the treatment of isolated conventional post-TxC for 6-8 months.

Study Sample Sample: All adult patients undergoing a heart transplant between January 2017 and December 2023 at Hospital de Messejana.

Inclusion Criteria Included: Patients of both sexes, aged ≥ 18 years, who have undergone heart transplantation between January 2017 and December 2023 and are under the care of the Heart Transplant and Heart Failure Unit at Hospital de Messejana.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes, aged ≥ 18 years, who have undergone heart transplantation between January 2017 and December 2023 and are under the care of the Heart Transplant and Heart Failure Unit at Hospital de Messejana.

Exclusion Criteria:

Patients who refuse to participate in the study, those with known hypersensitivity or intolerance to iSGLT2, individuals with type 1 diabetes mellitus, symptoms of hypotension, or systolic blood pressure below 80 mm Hg, an estimated glomerular filtration rate (eGFR) below 20 ml per minute per 1.73 m2 of body surface area, and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Allograft Vasculopathy | 6 to 8 months
  Cardiac Allograft Vasculopathy

SECONDARY OUTCOMES:
cardiovascular death | 6 to 8 months
  cardiovascular death
all-cause mortality | 6 to 8 months
  all-cause mortality
cardiovascular hospitalization | 6 to 8 months
  cardiovascular hospitalization
worsening glomerular filtration rate | 6 to 8 months
  sustained ≥50% decline in eGFR, occurrence of end-stage kidney disease or death due to kidney disease

OTHER OUTCOMES:
fasting glucose | 6 to 8 months
  fasting glucose
weight | 6 to 8 months
  weight
blood pressure | 6 to 8 months
  blood pressure
Rejection | 15 days post HTx
  Rejection in a subgroup of early post-Htx patients
urinary tract infection | 6 to 8 months
  urinary tract infection
Hypovolemia | 6 to 8 months
  Hypovolemia
limb amputation | 6 to 8 months
  limb amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Messejana Hospital, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided